CLINICAL TRIAL: NCT01982136
Title: Prospective Long-term Single Center Cohort Study Assessing Functional Outcome of Urethral Reconstructive Surgery
Brief Title: Functional Outcome of Urethral Reconstructive Surgery
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML9859; S55868 (Other: UZLeuven)
Record Dates: First submitted 2013-10-24; First posted 2013-11-13 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Urethral stricture: patients requiring surgery for urethral stricture
  Interventions: Procedure: end-to-end urethroplasty; Procedure: substitution urethroplasty (buccal mucosa); Procedure: substitution urethroplasty (pedicled skin flap)

INTERVENTIONS:
Procedure: end-to-end urethroplasty
Procedure: substitution urethroplasty (buccal mucosa)
Procedure: substitution urethroplasty (pedicled skin flap)

SUMMARY:
The analysis of the long-term outcomes and quality-of-life parameters after urethral reconstruction surgery.

DETAILED DESCRIPTION:
Urethroplasty is the surgical repair of a urethral stricture. Depending on the location, severity and length of the stricture, various techniques can be performed.

The first procedure consists of the excision of the stenotic segment and end-to-end anastomosis. Other procedures consist of widening the urethra with buccal mucosa as free graft or with vascularized (genital) skin flaps. The results of these techniques have been described in prospective cohort studies, but to date there is little good data about the functional outcome and quality-of-life with longer follow-up after this surgery.

The purpose of this study is to prospectively follow patients for functional outcome parameters and quality-of-life to obtain long-term information concerning these surgeries.

ELIGIBILITY:
Inclusion Criteria:

* male
* urethral stricture surgery
* informed consent

Exclusion Criteria:

* loss of follow-up
* not willing to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent urethral reconstruction in our center from 2009 to this date
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Quality Of Life: change from baseline (=preoperative value) | 6m, 1y, 2y, 3y, 4y
  Validated questionnaires (patient reported outcome measures) concerning general discomfort, micturition problems, erections, and the impact of those problems on their social life.
  * International Prostate Symptom Score - Quality of Life questionnaire (IPSS-QOL)
  * International Consultation of Incontinence - Lower Urinary Tract Symptoms Quality of Life questionnaire (ICIQ-LUTSQoL)

SECONDARY OUTCOMES:
Functional outcomes: micturition: change from baseline (=preoperative value) | 6m, 1y, 2y, 3y, 4y
  Validated questionnaires
  * International Consultation of Incontinence - Lower Urinary Tract Symptoms Quality of Life questionnaire (ICIQ-LUTSQoL)
  * Urogenital Distress Inventory short form (UDI-6)
Functional outcomes: erection: change from baseline (=preoperative value) | 6m, 1y, 2y, 3y, 4y
  Validated questionnaires
  * International Index of Erectile Dysfunction (IIEF)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Van der Aa, MD-PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium